CLINICAL TRIAL: NCT06398756
Title: The Impact of Aquatic Therapy on Walking, Balance Functions, and Quality of Life in Children With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Emel TURGUT VARAN, medical doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10026545
Record Dates: First submitted 2024-04-29; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Palsy
Keywords: aquatic therapy; rehabiltation
MeSH Terms: conditions — Cerebral Palsy | interventions — Aquatic Therapy

STUDY DESIGN:
Intervention Model Description: assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional rehabilitation (Active Comparator): 17 cerebral palsy patients will be included in the conventional rehabilitation program.
  Interventions: Other: conventional rehabilitation
- conventional rehabilitation and aquatic therapy (Active Comparator): 17 cerebral palsy patients will be included in the conventional rehabilitation and aquatic therapy program.
  Interventions: Other: aquatic therapy

INTERVENTIONS:
Other: conventional rehabilitation — 17 patients with cerebral palsy meeting the criteria will undergo conventional rehabilitation
  Arms: conventional rehabilitation
Other: aquatic therapy — 17 patients with cerebral palsy meeting the criteria will undergo convertional rehabilitation and aquatic therapy
  Arms: conventional rehabilitation and aquatic therapy

SUMMARY:
The purpose of the study is to contribute to the rehabilitation program by comparing the effects of traditional rehabilitation methods and aquatherapy given in addition to these methods in patients with cerebral palsy. If the superiority of the rehabilitation program including aquatherapy is demonstrated, evidence will be provided for its more widespread use.

DETAILED DESCRIPTION:
The participants will be divided into two groups as the study group and the control group. The study group will receive an aquatherapy rehabilitation program in addition to the conventional rehabilitation program, while the control group will only receive the conventional rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

1. Having a diagnosis of Hemiplegic Type or Diplegic Type Cerebral Palsy
2. Being between the ages of 3 and 16
3. Being at GMFCS levels I, II, and III
4. Having sufficient cognitive abilities such as understanding simple instructions, following them, and performing requested tasks
5. Parents and patients aged ≥ 9 agreeing to participate in the research

Exclusion Criteria:

1. Experiencing uncontrolled seizures
2. Having serious learning difficulties, behavioral problems, skin lesions, visual and/or hearing impairments that could affect function and participation
3. Active infection
4. Incontinence

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | baseline, after 1 month and 3 month changes.
  MAS 0: No increase in tone MAS 1: Minimal resistance or a catch and release at the end of the range of motion MAS 1+: Slight increase in tone, with minimal resistance felt in less than half of the range of motion MAS 2: Increased tone throughout most of the range of motion, but the joint can be easily moved MAS 3: Marked increase in tone, making passive movement difficult MAS 4: Rigidity in flexion or extension of the affected part
Gross Motor Function Measurement | baseline, after 1 month and 3 month changes.
  The Gross Motor Function Measurement (GMFM) is an assessment method used to determine the motor development level of children with cerebral palsy. Its purpose is to measure not just the quality of motor performance, but rather how much of the movement the child has accomplished.

SECONDARY OUTCOMES:
Pediatric Balance Scale | baseline, after 1 month and 3 month changes.
  The Pediatric Balance Scale (PBS)" is a functional balance measure that evaluates postural control while children perform activities they commonly engage in at home, school, and within the community. It consists of a 14-item scale, with each item scored from 0 to 4. The maximum score is 56.
The Functional Reach Test | baseline, after 1 month and 3 month changes.
  The Functional Reach Test is one of the dynamic balance assessment methods. It measures the maximum distance one can reach forward and sideways while standing upright.

CONTACTS AND LOCATIONS:
Overall Officials: Emel Turgut Varan, Medical Doctor, Principal Investigator — Ankara City Hospital Bilkent; Özlem Yılmaz Taşdelen, Professor Doctor, Study Director — Ankara City Hospital Bilkent; Evren Yaşar, Professor Doctor, Study Chair — Ankara City Hospital Bilkent; Hacer Han, Physical therapist, Study Chair — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital Physical Therapy and Rehabilitation Hospital, Ankara, Ankara, Bilkent-Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roostaei M, Baharlouei H, Azadi H, Fragala-Pinkham MA. Effects of Aquatic Intervention on Gross Motor Skills in Children with Cerebral Palsy: A Systematic Review. Phys Occup Ther Pediatr. 2017 Oct 20;37(5):496-515. doi: 10.1080/01942638.2016.1247938. Epub 2016 Dec 14. PMID 27967298